CLINICAL TRIAL: NCT01986374
Title: Intrauterine Injection of Human Chorionic Gonadotropin to Enhance Embryo Implantation
Brief Title: Injection of Hormone to Enhance Implantation in Embryo Transfer After IVF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servy Massey Fertility Insititute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCG 2013
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2013-11

CONDITIONS: Infertility
Keywords: IVF , embryo implantation, HCG
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HCG is introduced with small catheter. (Experimental): phase 1 non randomized pilot
  Interventions: Drug: HCG is introduced

INTERVENTIONS:
Drug: HCG is introduced — must have good blastocysts
  Other Names: Improve results of IVF and embryo transfer

SUMMARY:
The endometrium is deprived of signals form the embryo in IVF conditions. Studies suggest that placing HCG into the uterus prior to embryo transfer can enhance implantation.

DETAILED DESCRIPTION:
The study is in pilot phase, uncontrolled. The risks appear to be minimal and there are conflicting new reports being announced.

A small amount of fluid with HCG is injected into the uterus. HCG is a potent signal to the uterus for preparation for implantation.

This is not a funded study. Three published studies suggest the approach is valid; one refutes the concept.

ELIGIBILITY:
Inclusion Criteria:

- infertility patients undergoing IVF with good expectation of two embryos day 3 or day 5. must speak and read English. Includes donor eggs.

Exclusion Criteria:abnormal uterus

-

Ages: 21 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
HCG enhances pregnancy rate | 9 months.
  compare pregnancy rates to established clinical norms.

SECONDARY OUTCOMES:
implantation rate | 18 months
  compare implantation rate per embryo to clinical norms.
ongoing pregnancy rate | 22 months
  compare success to clinical norms

CONTACTS AND LOCATIONS:
Overall Officials: Joe B Massey, MD, Study Chair — Servy Massey Fertilty Institute
Locations (1):
- Servy Massey Fertility Insititute, Atlanta, Georgia, United States

REFERENCES:
- [Background] Mansour R, Tawab N, Kamal O, El-Faissal Y, Serour A, Aboulghar M, Serour G. Intrauterine injection of human chorionic gonadotropin before embryo transfer significantly improves the implantation and pregnancy rates in in vitro fertilization/intracytoplasmic sperm injection: a prospective randomized study. Fertil Steril. 2011 Dec;96(6):1370-1374.e1. doi: 10.1016/j.fertnstert.2011.09.044. Epub 2011 Nov 1. PMID 22047664
- [Background] Zarei A, Parsanezhad ME, Younesi M, Alborzi S, Zolghadri J, Samsami A, Amooee S, Aramesh S. Intrauterine administration of recombinant human chorionic gonadotropin before embryo transfer on outcome of in vitro fertilization/ intracytoplasmic sperm injection: A randomized clinical trial. Iran J Reprod Med. 2014 Jan;12(1):1-6. PMID 24799855
- [Background] Santibanez A, Garcia J, Pashkova O, Colin O, Castellanos G, Sanchez AP, De la Jara JF. Effect of intrauterine injection of human chorionic gonadotropin before embryo transfer on clinical pregnancy rates from in vitro fertilisation cycles: a prospective study. Reprod Biol Endocrinol. 2014 Jan 29;12:9. doi: 10.1186/1477-7827-12-9. PMID 24476536
- [Background] Hong KH, Forman EJ, Werner MD, Upham KM, Gumeny CL, Winslow AD, Kim TJ, Scott RT Jr. Endometrial infusion of human chorionic gonadotropin at the time of blastocyst embryo transfer does not impact clinical outcomes: a randomized, double-blind, placebo-controlled trial. Fertil Steril. 2014 Dec;102(6):1591-5.e2. doi: 10.1016/j.fertnstert.2014.08.006. Epub 2014 Sep 16. PMID 25234040